CLINICAL TRIAL: NCT02041455
Title: Phase II Role of Immune-pineal Axis in Fibromyalgia: Noradrenergic Modulation and Chronotherapeutic Aspects
Brief Title: Immune-Pineal Axis Function in Fibromyalgia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-261
Record Dates: First submitted 2014-01-16; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Melatonin; Amitriptylin; Imune-pineal axis
MeSH Terms: conditions — Fibromyalgia | interventions — Melatonin; Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Melatonin and Placebo (Experimental): Melatonin 10mg and placebo, once in the evening, for 6 weeks.
  Interventions: Drug: Melatonin and Placebo
- Amitriptyline and placebo (Experimental): Amitriptyline 25mg and placebo, once in the evening, for 6 weeks.
  Interventions: Drug: Amitriptyline and Placebo
- Melatonin and Amitriptylin (Active Comparator): Melatonin 10mg and Amitriptylin 25mg, once in the evening, for 6 weeks.
  Interventions: Drug: Melatonin and Amitriptylin

INTERVENTIONS:
Drug: Melatonin and Placebo
  Arms: Melatonin and Placebo
Drug: Amitriptyline and Placebo
  Arms: Amitriptyline and placebo
Drug: Melatonin and Amitriptylin
  Arms: Melatonin and Amitriptylin

SUMMARY:
Fibromyalgia is a common condition in clinical medical practice, characterized by diffuse musculoskeletal pain. Sleep disorders, chronic fatigue, depression, intestinal disorders and headache are also commonly associated with the syndrome .

Although the etiology of this syndrome is not well defined yet, it means involve multiple mechanisms, including low levels of serotonin, increased substance P in cerebrospinal fluid and altered circadian variation in sympathetic - parasympathetic balance, consistent with changes in sympathetic hyperactivity at night .

The immune - pineal system, formed by the integration of the adrenergic and immune systems pineal gland, appears to be involved in the genesis of the dysfunctions found in fibromyalgia. Melatonin is secreted by the pineal gland and has promoter activity of sleep. Studies show that melatonin and its precursors , serotonin and tryptophan are reduced in patients with fibromyalgia.

The present study aims to evaluate the relationship of immune - pineal system in the process of fibromyalgia , since dysfunction of this axis appears to govern the cascading events that participate in the pathophysiological process of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-65 years old
* Fibromyalgia according to the criteria of the American College of Rheumatology (Wolfe 2010)
* Sign the informed consent
* Patients can take medication for chronic pain ( antidepressants , antiepileptics, for example), since there are at least two months

Exclusion criteria:

* patients who did not understand the Portuguese
* diagnosis of malignancies, severe psychiatric disorders , sleep disorders not related to fibromyalgia (apnea , sleepwalking , restless leg syndrome), Alzheimer's disease or any disease (rheumatologic, neurological, etc.) that can modify the evaluations or outcomes
* alcohol abuse or drug addiction
* patients who are performing acupuncture
* BMI greater than 35 ( BMI = body mass index) .
* Patients with history of allergy to amitriptyline or/and melatonin or any other contraindication for the use of these drugs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in pain on Fibromyalgia Impact Questionnaire (FIQ) at week 6 | Baseline, week 6
Change from Baseline in Pain Pressure Threshold (PPT) at week 6 | Baseline, week 6
  Pain Pressure Threshold by Fischer algometer on the tender points.
Change from Baseline Brain-derived neurotrophic factor at week 6 | Baseline, week 6

SECONDARY OUTCOMES:
Change from Baseline of the Pittsburgh Sleep Quality Index (PSQI) at week 6 | Baseline, week 6
Change from Baseline of the Pain Catastrophizing Scale at week 6 | Baseline; week 6
  Catastrophic thinking related to pain

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei d Caumo, PhD, Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] de Zanette SA, Vercelino R, Laste G, Rozisky JR, Schwertner A, Machado CB, Xavier F, de Souza IC, Deitos A, Torres IL, Caumo W. Melatonin analgesia is associated with improvement of the descending endogenous pain-modulating system in fibromyalgia: a phase II, randomized, double-dummy, controlled trial. BMC Pharmacol Toxicol. 2014 Jul 23;15:40. doi: 10.1186/2050-6511-15-40. PMID 25052847